CLINICAL TRIAL: NCT03119779
Title: The Effect of Pulpotomy (Partial or Complete) Using Resin-Modified Calcium Silicate Versus MTA-Anglus on Survival Rate of Cariously-Exposed Vital Young Permanent Molars:A Randomized Clinical Trial
Brief Title: Effect of Pulpotomy Using TheraCal Versus MTA on Survival Rate of Cariously-Exposed Vital Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Passant Nagy, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBD-CU-2014-09-15
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Caries, Dental
Keywords: pulpotomy; deep caries; permanent molars; MTA
MeSH Terms: conditions — Dental Caries | interventions — TheraCal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TheraCal vital pulp therapy (Experimental): Using rubber dam isolation we will remove the caries using large round but under copious amount of coolant and if carious exposure occur, part of the pulp chamber will be removed using sharp spoon excavator. After complete removal of the caries and control of bleeding, then direct application of incremental layers of TheraCal using the tip of the syringe container of the material and each layer should not exceed 1 mm then light curing each increment. Then Riva self-cure glass-ionomer base and composite resin final restoration. We will take immediate standardized postoperative periapical radiographs.
  Interventions: Drug: TheraCal
- MTA vital pulp therapy (Active Comparator): Using rubber dam isolation we will remove the caries using large round but under copious amount of coolant and if carious exposure occur, part of the pulp chamber will be removed using sharp spoon excavator. After complete removal of the caries and control of bleeding, then direct application of freshly mixed MTA-Anglus on sterile glass slap. MTA application then gentle condensation over wet cotton till MTA thickness is about 2-3 mm thickness and removal of excess material from walls of pulp chamber. Application of wet cotton for 15 min. to achieve initial setting of MTA. Then Riva self-cure glass-ionomer base and composite resin final restoration. We will take immediate standardized postoperative periapical radiographs.
  Interventions: Drug: MTA-Anglus

INTERVENTIONS:
Drug: MTA-Anglus — MTA-Anglus freshly mixed according to manufacturer instructions over glass slap and applied to pulp stump and application of wet cotton for 15 min. till initial setting occur.
  Other Names: MTA-Anglus vital pulp therapy
  Arms: MTA vital pulp therapy
Drug: TheraCal — TheraCal directly applied from the syringe container tip to pulp stump over incremental layers each layer should not exceed 1 mm thickness and each layer will be light cured for 20 sec.
  Other Names: TheraCal vital pulp therapy
  Arms: TheraCal vital pulp therapy

SUMMARY:
Objective:

To assess which is the most efficient pulpotomy medicament on tooth survival in patients with a cariously-exposed vital young permanent molar regarding: absence of postoperative pain, sinus or swelling, internal/ external root resorption, periapical radiolucency), root maturation and decrease chair side time of treated patient.

Trial design Randomized Clinical Trial (RCT), double-blinded with parallel group and allocation ratio (1:1), equivalence framework.

DETAILED DESCRIPTION:
Preoperative records will be taken (photos, conventional periapical radiographs, and impression to construct acrylic stent to help standardization on follow up apical radiographs). Administration of inferior alveolar nerve block then using rubber dam isolation one of the investigators will remove the caries using large round but under copious amount of coolant and if carious exposure occur, part of the pulp chamber will be removed using sharp spoon excavator. Then the pulp status will be assessed if bleeding is controlled with direct irrigation with distilled water for 2 minutes then next step will be taken but if not continue excavation of the pulp till bleeding is controlled. if bleeding is not controlled after performing complete pulpotomy, tooth will be excluded from the study Then direct application of capping materials (TheraCal or MTA) according to manufacturer instructions, then Riva self-cure glass-ionomer base and composite resin final restoration. One of the investigators will take immediate standardized postoperative periapical radiographs. Follow-up will be for 12 months. Pre-calibrated blinded dentists will assess out comes separately.

ELIGIBILITY:
Inclusion Criteria:

* Restorable permanent molars with deep caries and pain could be relieved with analgesics

Exclusion Criteria:

* criteria of exclusion of teeth were:

  * pathological mobility, swelling or tenderness to percussion/palpation;
  * pathology is shown in the pre-operative radiographic as resorption periradicular or furcation radiolucency, or a widened periodontal ligament space;
  * at the operative procedure, hemorrhage control is unachievable

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Survival rate | 12 months
  absence of any complication or complementary treatment (absence of spontaneous pain or swelling)

SECONDARY OUTCOMES:
periapical radiolucency | 12 months
  presence or absence of periapical radiolucency radiographically
internal/ external root resorption | 12 months
  presence or absence of internal/ external root resorption radiographically
Root maturation | 12 months
  Root maturation assessment radiographically

OTHER OUTCOMES:
Time lapse till final restoration performed | from 5 till 20 minutes
  measured using stop watch to assess which material needs less chair side time to be finished.

CONTACTS AND LOCATIONS:
Overall Officials: Passant Nagi, MSc, Principal Investigator — Assisternt lecturer

IPD SHARING:
Plan to Share IPD: No